CLINICAL TRIAL: NCT01892358
Title: Preventing Bacterial and Viral Infections Among Injection Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA034957; 1210-003 (Other: Butler Hospital)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Bacterial Infection; HIV
Keywords: injection drug use
MeSH Terms: conditions — Bacterial Infections | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SKIN Intervention (Active Comparator): Participants will receive the SKIN intervention at Baseline and 1-mo interviews.
  Interventions: Behavioral: SKIN Intervention
- Assessment-Only (Placebo Comparator): Participants in this arm will receive treatment-as-usual
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: SKIN Intervention
  Arms: SKIN Intervention
Other: Treatment as Usual
  Arms: Assessment-Only

SUMMARY:
We propose a randomized controlled trial (RCT) of the Skin intervention, compared to an assessment-only condition (both groups receive rapid HIV testing, a review of testing results, and brief HIV prevention counseling) among 350 injection drug users recruited during an acute medical hospitalization at Boston Medical Center. In the general hospital setting, injection drug users who otherwise might not seek care are accessible and teachable, and the presence of a drug-related illness can set the stage for patients to be more receptive to interventions2. We hypothesize that the Skin intervention will produce better outcomes at 1-, 3-, 6-, 9-, and 12-month(s) post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* report injection of heroin, cocaine, or methamphetamine (meth) on at least three different days in the week prior to admission
* have injected heroin, cocaine, or meth for at least three months
* positive urine screen for heroin, cocaine, or meth

Exclusion Criteria:

* currently psychotic (e.g., responding to internal stimuli through observed hallucinations or delusions), homicidal or suicidal
* cannot provide informed consent
* not able to complete interviews in English (expected to exclude <5% of IDUs)
* in police custody, expecting incarceration
* unable to provide names and contact information for at least two verifiable locator persons who will know where to find them for retention/follow-up purposes
* plan to move out of the Boston area in the next 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2013-09; Primary Completion 2019-08 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
bacterial infections | one year
high-risk behavior | one year
health service use | one year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Freibott CE, Phillips KT, Anderson BJ, Stewart C, Liebschutz JM, Stein MD. Under the Skin: The Relationship Between Subcutaneous Injection and Skin Infections Among People Who Inject Drugs. J Addict Med. 2022 Mar-Apr 01;16(2):164-168. doi: 10.1097/ADM.0000000000000844. PMID 33813580
- [Derived] Stein MD, Phillips KT, Herman DS, Keosaian J, Stewart C, Anderson BJ, Weinstein Z, Liebschutz J. Skin-cleaning among hospitalized people who inject drugs: a randomized controlled trial. Addiction. 2021 May;116(5):1122-1130. doi: 10.1111/add.15236. Epub 2020 Sep 21. PMID 32830383